CLINICAL TRIAL: NCT03271866
Title: The Effect of Metformin Treatment on Cognitive Impairment in Patients With Schizophrenia Co-morbid Metabolic Syndrome: a Prospective Cohort Study
Brief Title: Metformin Treatment on Cognitive Impairment of Schizophrenia Co-morbid Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Renrong Wu, Professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WU201708MET
Record Dates: First submitted 2017-08-30; First posted 2017-09-05 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Metabolic syndrome; Metformin; Cognitive impairment; Clinical trial
MeSH Terms: conditions — Schizophrenia; Metabolic Syndrome; Cognitive Dysfunction | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Two groups were observed longitudinally for 24 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- metformin treatment (Other)
  Interventions: Drug: metformin
- non-metformin treatment (No Intervention)

INTERVENTIONS:
Drug: metformin — metformin 1500mg per day
  Arms: metformin treatment

SUMMARY:
In this study, the investigators will investigate the impact and the related mechanism of metformin treatment on cognitive impairment of schizophrenia with a high risk of metabolic syndrome. Patients will be randomized to the metformin group or non-metformin control group (40 patients per arm) for 24 weeks. Clinical assessment will be done at screen/baseline, 4 weeks, 12 weeks, and 24 weeks. The specific aims are to compare the metformin group versus controls on 1) clinical core symptoms; 2) cognition. Biological samples also will be collected, and stored to research related mechanisms.

DETAILED DESCRIPTION:
In this study, the investigators will investigate the impact and the related mechanism of metformin treatment on cognitive impairment of schizophrenia with a high risk of metabolic syndrome. Patients will be randomized to the metformin group or non-metformin control group (40 patients per arm) . Clinical assessment will be done at screen/baseline, 4 week, 12 week and 24 week. The specific aims are to compare the metformin group versus controls on: 1) clinical core symptoms; 2) cognition. Biological samples also will be collected, and stored to research related mechanisms. Clinical symptoms will be measured by the Positive and Negative Syndrome Scale and Calgary Depression Scale for Schizophrenia (Chinese version). Cognitive function will be assessed by the MATRICS Consensus Cognitive Battery.

The investigators hypothesize that 1) metformin may improve the cognitive impairment of schizophrenia patients; 2) metformin may alter oxidative stress indexes or inflammatory biomarkers thus influencing the oxidative and inflammatory mechanism, and the structure and function of the hippocampus that may be significantly associated with cognitive function.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the Diagnostic and Statistical Manual (DSM-5) diagnostic criteria for schizophrenia;
2. Duration of illness less than 5 years with current symptoms exacerbation;
3. Male and female aged 18 to 65 years;
4. PANSS total score < 60 and CDSS-C total score < 6;
5. Signed the study consent for participation;
6. Patients with higher risk factors for MetS, or patients who gained weight > 10% of their pre-drug weight within the first year after antipsychotic medication.

Exclusion Criteria:

1. Having a history of substance dependence or abuse or whose symptoms are caused by other diagnosable mental disorders;
2. Having a history of traumatic brain injury, seizures, or other known neurological or organic diseases of the central nervous system;
3. Taking antidepressants, stimulants, mood stabilizers or accepting electricity shock treatment;
4. Having current suicidal or homicidal thoughts or any safety concern by research staff that cannot be managed in an inpatient setting;
5. The routine blood tests showing abnormal renal, and liver function;
6. Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-08-28 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive improvement will be assessed using the MATRICS Consensus Cognitive Battery (MCCB) composite score | 12 weeks
  The investigators will use the MATRICS Consensus Cognitive Battery (MCCB) Composite score as primary cognitive outcome measure before and after treatment at different follow up point.

SECONDARY OUTCOMES:
Change of clinical symptoms by PANSS | 12 weeks
  The change of Positive And Negative Syndrome Scale (PANSS) total, positive and negative symptoms before and after treatment at different follow up point.

OTHER OUTCOMES:
Depression by CDSS-C | 12 weeks
  The investigators will assess depression by Calgary Depression Scale for Schizophrenia （Chinese version, CDSS-C）
Biological markers will be measured by ELISA | 12 weeks
  The oxidative stress indexes and inflammatory biomarkers will measured by Enzyme-linked Immuno Sorbent Assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Tiannan Shao, M.D., Ph.D., Principal Investigator — Central South University; Dongyu Kang, M.D., Principal Investigator — Central South University; Renrong Wu, M.D., Ph.D., Study Chair — Central South University
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

REFERENCES:
- [Background] Lindenmayer JP, Khan A, Kaushik S, Thanju A, Praveen R, Hoffman L, Cherath L, Valdez G, Wance D. Relationship between metabolic syndrome and cognition in patients with schizophrenia. Schizophr Res. 2012 Dec;142(1-3):171-6. doi: 10.1016/j.schres.2012.09.019. Epub 2012 Oct 26. PMID 23106932
- [Background] Bora E, Akdede BB, Alptekin K. The relationship between cognitive impairment in schizophrenia and metabolic syndrome: a systematic review and meta-analysis. Psychol Med. 2017 Apr;47(6):1030-1040. doi: 10.1017/S0033291716003366. Epub 2016 Dec 29. PMID 28032535
- [Background] Ying MA, Maruschak N, Mansur R, Carvalho AF, Cha DS, McIntyre RS. Metformin: repurposing opportunities for cognitive and mood dysfunction. CNS Neurol Disord Drug Targets. 2014;13(10):1836-45. doi: 10.2174/1871527313666141130205514. PMID 25470390
- [Derived] Cai J, Xiao J, Long Y, Cao T, Lin C, Hei G, Wang W, Kang D, Huang J, Shao T, Cai H, Wu R. Metformin-improved cognitive impairment in patients with schizophrenia is correlated with activation of tricarboxylic acid cycle and restored functional connectivity of hippocampus. BMC Med. 2025 Jul 1;23(1):349. doi: 10.1186/s12916-025-04218-4. PMID 40597190
- [Derived] Shao T, Huang J, Zhao Y, Wang W, Tian X, Hei G, Kang D, Gao Y, Liu F, Zhao J, Liu B, Yuan TF, Wu R. Metformin improves cognitive impairment in patients with schizophrenia: associated with enhanced functional connectivity of dorsolateral prefrontal cortex. Transl Psychiatry. 2023 Oct 11;13(1):315. doi: 10.1038/s41398-023-02616-x. PMID 37821461